CLINICAL TRIAL: NCT06250361
Title: Identification of Factors ASsociaTed With a Delayed Diagnosis in Crohn's Disease: the FAST Study
Brief Title: Identification of Factors ASsociaTed With a Delayed Diagnosis in Crohn's Disease
Acronym: FAST
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Responsible Party: Sponsor
Other Study IDs: GETAID-2023-01
Record Dates: First submitted 2024-01-15; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-01

CONDITIONS: Crohn Disease
Keywords: IBD; CROHN; CD
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire completion — A questionnaire will be completed by the participant and their gastroenterologist. Estimated completion time is 30 minutes for the patient, 10 minutes for the gastroenterologist.

SUMMARY:
The goal of this observational study is to determine the factors associated with a delayed diagnosis and/or an immediately complicated disease for CD patients.

A questionnaire will be completed by the patients, each questionnaire has a patient section and a physician section.

DETAILED DESCRIPTION:
Number of patients expected : at least 600, coming from all types of practices (ANGH (expert hospitals), GETAID (expert university hospitals) and CREGG (expert private practice)).

Recruitment period : 1 year

Primary endpoint : The primary endpoint is the description of the factors linked to:

* The IBD
* The patient (see patient questionnaire in annex 1)
* The health care system
* The patient's self-care

Secondary endpoint :

* Validation of the "red flags" in a prospective cohort.
* Comparison with the EPIMAD population, especially the location and severity.

ELIGIBILITY:
Inclusion Criteria:

* Crohn's disease diagnosed less than a year prior to inclusion
* Written consent
* Age ≥ 18 years

Exclusion Criteria:

* Diagnosis of Crohn's disease more than one year before inclusion
* Patient protected by the law
* Patient without health cover

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Crohn's disease, going to ANGH (expert hospitals), GETAID (expert university hospitals) and CREGG (expert private practice) centres, who have been diagnosed within the year before the inclusion visit.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Number of patient's visits to doctors between the appearance of the first symptoms and the diagnosis of the disease. | Day 1 from appearence of first symptoms and the diagnosis of the disease.
  Number of patient's visits to doctors between the appearance of the first symptoms and the diagnosis of the disease.
Number of exams performed between the appearance of the first symptoms and the diagnosis of the disease. | Day 1 from appearence of first symptoms and the diagnosis of the disease.
  Number of exams performed between the appearance of the first symptoms and the diagnosis of the disease.
Number of medical specialties consulted between the appearance of the first symptoms and the diagnosis of the disease. | Day 1 from appearence of first symptoms and the diagnosis of the disease.
  Number of medical specialties consulted between the appearance of the first symptoms and the diagnosis of the disease.

SECONDARY OUTCOMES:
Number of predictive factors associated with a delayed diagnosis | Day 1
  Number of predictive factors associated with a delayed diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane Nahon, PhD, Principal Investigator — Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives

IPD SHARING:
Plan to Share IPD: No